CLINICAL TRIAL: NCT00122863
Title: Duloxetine 60 to 120 mg Once Daily Compared With Placebo in the Prevention of Relapse in Generalized Anxiety Disorder
Brief Title: Duloxetine Compared With Placebo in the Prevention of Relapse in Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7108; F1J-MC-HMDV
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride
Drug: placebo

SUMMARY:
This is a clinical trial assessing the time to relapse of anxiety symptoms among patients with generalized anxiety disorder who have responded to duloxetine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with generalized anxiety disorder (GAD) in the absence of major depressive disorder (MDD). Patients must suffer from GAD and not from an adjustment disorder or anxiety disorder not otherwise specified (NOS). Symptoms of GAD should not be situational in nature.

Exclusion Criteria:

* Any current and primary diagnosis other than GAD. Patients diagnosed with or who have a history of MDD within the past 6 months OR patients diagnosed with or who have a history of panic disorder, post-traumatic stress disorder (PTSD), or an eating disorder within the past year OR patients who have been diagnosed with obsessive- compulsive disorder (OCD), bipolar affective disorder, psychosis, factitious disorder or somatoform disorders during their lifetime.
* History of alcohol or any psychoactive substance abuse of dependence (as defined in the DSM-IV-TR) within the past 6 months
* Serious medical illness, including cardiovascular, hepatic, renal, respiratory, hematologic, endocrinologic, or neurologic disease, or clinically significant laboratory abnormality that is not stabilized or is anticipated to require hospitalization within 6 months, in the opinion of the investigator. Clinically significant laboratory abnormalities are those, that, in the judgement of the investigator, indicate a serious medical problem.
* Acute liver injury (such as hepatitis) or severe cirrhosis (Child- Pugh Class C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2005-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Assess the long-term maintenance of efficacy of duloxetine 60 to 120 mg QD compared with placebo by a comparison of the time to relapse among patients with GAD who responded to duloxetine during the open-label acute therapy phase after 22 to 26 weeks.

SECONDARY OUTCOMES:
Self-reported anxiety symptomatology
Pain
Quality of Life
Clinical Global Improvement and HAMA Factor scores
Maintenance of Effect

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (47):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Charles, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita Falls, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodstock, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- France (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aix-en-Provence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arcachon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bourg-des-Comptes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clermont-Ferrand
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montigny-lès-Metz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mulhouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orvault
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hildesheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Werneck
- Netherlands (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Almere Stad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijverdal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
- Portugal (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce

REFERENCES:
- [Derived] Perlis RH, Fijal B, Dharia S, Houston JP. Pharmacogenetic investigation of response to duloxetine treatment in generalized anxiety disorder. Pharmacogenomics J. 2013 Jun;13(3):280-5. doi: 10.1038/tpj.2011.62. Epub 2012 Jan 17. PMID 22249355
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com